CLINICAL TRIAL: NCT02935738
Title: Improvement in Pregnancy Outcomes in Immunologically Infertile Male Patients Undergoing Prednisolone Treatment and Conventional IVF Preceded by Sperm Penetration Assay: A Randomized Controlled Trial
Brief Title: Prednisolone Improves IVF Outcomes in Men With Anti-sperm Antibodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barz IVF Center for Infertility Treatment and Embryo Research (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prednisolone-SPA-IVF
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Reproductive Sterility
Keywords: prednisolone; anti-sperm antibodies; sperm penetration assay
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prednisolone treated men / positive SPA / IVF (Experimental): Infertile men, with anti-sperm antibodies, were treated with prednisolone tablet, which is an intermediate acting corticosteroid, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was started with a dose of 5mg, tid, for two weeks followed by 5mg bid for five days. This was further tapered to one tablet of 5mg/day for two days. Patients were then given one week of rest from the treatment, before this prednisolone regimen was repeated for another two cycles. Prednisolone treated men, who recovered from anti-sperm antibodies, underwent then sperm penetration assay (SPA) using zona-free hamster ova. Couples with male partners having positive SPA results (greater than five) were admitted to conventional in vitro fertilization (IVF) cycles.
  Interventions: Drug: Prednisolone treatment
- Prednisolone treated men / negative SPA / ICSI (Experimental): Infertile men, with anti-sperm antibodies, were treated with prednisolone tablet, which is an intermediate acting corticosteroid, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was started with a dose of 5mg, tid, for two weeks followed by 5mg bid for five days. This was further tapered to one tablet of 5mg/day for two days. Patients were then given one week of rest from the treatment, before this prednisolone regimen was repeated for another two cycles. Prednisolone treated men, who recovered from anti-sperm antibodies, underwent then sperm penetration assay (SPA) using zona-free hamster ova. Couples with male partners having negative SPA results (equal or less than five) were admitted to intracytoplasmic sperm injection (ICSI) cycles.
  Interventions: Drug: Prednisolone treatment
- Control men / positive SPA / IVF (No Intervention): Infertile men with anti-sperm antibodies who were not treated with prednisolone, which is an intermediate acting corticosteroid, underwent sperm penetration assay (SPA) using zona-free hamster ova. Couples with male partners having positive SPA results (more than five) were then admitted to in vitro fertilization (IVF) cycle.
- Control men / negative SPA / ICSI (No Intervention): Infertile men with anti-sperm antibodies who were not treated with prednisolone, which is an intermediate acting corticosteroid, underwent sperm penetration assay (SPA) using zona-free hamster ova. Couples with male partners having negative SPA results (equal or less than five) were then admitted to intracytoplasmic sperm injection (ICSI) cycles.

INTERVENTIONS:
Drug: Prednisolone treatment — Infertile men were treated with prednisolone tablet, which is an intermediate acting corticosteroid, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was started with a dose of 5mg, tid, for two weeks followed by 5mg bid for five days. This was further tapered to one tablet of 5mg/day for two days. Patients were then given one week of rest from the treatment, before this prednisolone regimen was repeated for another two cycles.
  Other Names: Experimental
  Arms: Prednisolone treated men / negative SPA / ICSI; Prednisolone treated men / positive SPA / IVF

SUMMARY:
Corticosteroids have been indicated to treat men with ASAs. Although many studies have confirmed the clinical therapeutic significance of corticosteroids in the treatment of men with ASAs, other studies have not found a therapeutic significance for corticosteroids in the treatment of men with ASAs. Moreover, although some reports have shown high fertilization and conception rates in couples when husbands did not have ASAs, other reports have shown that ASAs do not have a negative effect on fertilization and conception rates. These contradictory results have left the therapeutic effect of corticosteroids in men with ASA in continuing controversy. This controversy is also extended to include the usefulness of assisted reproductive technology (ART) in the treatment of patients with ASAs. In this regard, although some studies have shown that the pregnancy rate following in vitro fertilization (IVF) or intracellular sperm injection (ICSI) were similar in men with or without ASA or did not associate with ASA, others reported the superiority of ICSI over IVF and intrauterine insemination over natural intercourse in men with ASAs. It is possible that some patients with ASAs also have an additional problem(s) related to sperm binding to the oolemma and fusion into the ovum as well as sperm head decondensation. The latter condition may negatively influence or mask the clinical significance of corticosteroids on pregnancy rates in patients with ASAs. Some patients might not have benefited from corticosteroids and conventional IVF treatments due to the impaired sperm fusogenic capacity in addition to ASAs. Human sperm penetration assay (SPA), of the hamster oocyte free from zona pellucida, is a sensitive tool that can address such potential impairment of sperm binding with the oolemma and fusion into the oocyte as well as sperm head decondensation. Males with poor SPA results benefit from ICSI whereas those with good SPA results can still benefit from conventional IVF.

The present study was therefore conducted to address the therapeutic usefulness of a corticosteroid named prednisolone in the treatment of immunologically infertile men undergoing IVF or ICSI determined by SPA.

DETAILED DESCRIPTION:
This prospective study was conducted at the Barz IVF Center for Infertility Treatment and Embryo Research, Erbil, Kurdistan Region, Iraq and the Baghdad University Teaching Hospital of the College of Medicine, University of Baghdad, Baghdad, Iraq between October 2014 and May 2016. In all cases, the wife's ova were inseminated with the husband's semen samples. Identified men with positive ASAs were randomly assigned for treatment with or without prednisolone for three cycles. Infertile men were treated with prednisolone tablet, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was started with a dose of 5mg, tid, for two weeks followed by 5mg bid for five days. This was further tapered to one tablet of 5mg/day for two days. Patients were then given one week of rest from the treatment, before this prednisolone regimen was repeated for another two cycles

Treated men that recovered from ASAs and control patients underwent SPA. Patients with positive or negative SPA results were then admitted to conventional IVF or ICSI cycles, respectively. Only the first embryo transfer cycle following IVF or ICSI was included in this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female partners had complete or partial tubal patency
* Male partners with anti-sperm antibodies
* Male partners with sperm count > 35 million/ml.

Exclusion Criteria:

* Female partners with polycystic ovary
* Female partners with endometriosis
* Female partners with abnormal profile of reproductive hormones
* Female partners with abnormal profile of thyroid hormones
* Male partners with seminal fluid infections (e.g. leukospermia)
* Male partners with abnormal profile of reproductive hormones
* Male partners with abnormal profile of thyroid hormones

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saeeda A. Muhsen, DVM, PhD, Principal Investigator — Barz IVF Center for Infertility Treatment and Embryo Research

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Omu AE, al-Qattan F, Abdul Hamada B. Effect of low dose continuous corticosteroid therapy in men with antisperm antibodies on spermatozoal quality and conception rate. Eur J Obstet Gynecol Reprod Biol. 1996 Nov;69(2):129-34. doi: 10.1016/0301-2115(95)02539-1. PMID 8902446
- [Background] Hendry WF, Treehuba K, Hughes L, Stedronska J, Parslow JM, Wass JA, Besser GM. Cyclic prednisolone therapy for male infertility associated with autoantibodies to spermatozoa. Fertil Steril. 1986 Feb;45(2):249-54. doi: 10.1016/s0015-0282(16)49163-6. PMID 3949025
- [Background] Hendry WF, Hughes L, Scammell G, Pryor JP, Hargreave TB. Comparison of prednisolone and placebo in subfertile men with antibodies to spermatozoa. Lancet. 1990 Jan 13;335(8681):85-8. doi: 10.1016/0140-6736(90)90548-j. PMID 1967425
- [Background] Keane D, Jenkins DM, Higgins T, O'Neill M, Mulcahy MF, Ferriss JB. The effect of intermittent steroid therapy on anti-sperm antibody levels. Eur J Obstet Gynecol Reprod Biol. 1995 Nov;63(1):75-9. doi: 10.1016/0301-2115(95)02217-u. PMID 8674571
- [Background] Bals-Pratsch M, Doren M, Karbowski B, Schneider HP, Nieschlag E. Cyclic corticosteroid immunosuppression is unsuccessful in the treatment of sperm antibody-related male infertility: a controlled study. Hum Reprod. 1992 Jan;7(1):99-104. doi: 10.1093/oxfordjournals.humrep.a137568. PMID 1551969
- [Background] De Almeida M, Feneux D, Rigaud C, Jouannet P. Steroid therapy for male infertility associated with antisperm antibodies. Results of a small randomized clinical trial. Int J Androl. 1985 Apr;8(2):111-7. doi: 10.1111/j.1365-2605.1985.tb00824.x. PMID 3894245
- [Background] Haas GG Jr, Manganiello P. A double-blind, placebo-controlled study of the use of methylprednisolone in infertile men with sperm-associated immunoglobulins. Fertil Steril. 1987 Feb;47(2):295-301. PMID 3545909
- [Background] Vazquez-Levin MH, Notrica JA, Polak de Fried E. Male immunologic infertility: sperm performance on in vitro fertilization. Fertil Steril. 1997 Oct;68(4):675-81. doi: 10.1016/s0015-0282(97)00255-0. PMID 9341610
- [Background] Ayvaliotis B, Bronson R, Rosenfeld D, Cooper G. Conception rates in couples where autoimmunity to sperm is detected. Fertil Steril. 1985 May;43(5):739-42. doi: 10.1016/s0015-0282(16)48557-2. PMID 3996618
- [Background] Pagidas K, Hemmings R, Falcone T, Miron P. The effect of antisperm autoantibodies in male or female partners undergoing in vitro fertilization-embryo transfer. Fertil Steril. 1994 Aug;62(2):363-9. doi: 10.1016/s0015-0282(16)56892-7. PMID 8034086
- [Background] Zini A, Lefebvre J, Kornitzer G, Bissonnette F, Kadoch IJ, Dean N, Phillips S. Anti-sperm antibody levels are not related to fertilization or pregnancy rates after IVF or IVF/ICSI. J Reprod Immunol. 2011 Jan;88(1):80-4. doi: 10.1016/j.jri.2010.09.002. Epub 2010 Dec 15. PMID 21111486
- [Background] Zini A, Fahmy N, Belzile E, Ciampi A, Al-Hathal N, Kotb A. Antisperm antibodies are not associated with pregnancy rates after IVF and ICSI: systematic review and meta-analysis. Hum Reprod. 2011 Jun;26(6):1288-95. doi: 10.1093/humrep/der074. Epub 2011 Mar 23. PMID 21429953
- [Background] Lahteenmaki A, Reima I, Hovatta O. Treatment of severe male immunological infertility by intracytoplasmic sperm injection. Hum Reprod. 1995 Nov;10(11):2824-8. doi: 10.1093/oxfordjournals.humrep.a135800. PMID 8747025
- [Background] Robinson JN, Forman RG, Nicholson SC, Maciocia LR, Barlow DH. A comparison of intrauterine insemination in superovulated cycles to intercourse in couples where the male is receiving steroids for the treatment of autoimmune infertility. Fertil Steril. 1995 Jun;63(6):1260-6. doi: 10.1016/s0015-0282(16)57608-0. PMID 7750598

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisolone Treated Men / Negative SPA / ICSI: Infertile men, with anti-sperm antibodies, were treated with prednisolone tablet, which is an intermediate acting corticosteroid, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was started with a dose of 5mg, tid, for two weeks followed by 5mg bid for five days. This was further tapered to one tablet of 5mg/day for two days. Patients were then given one week of rest from the treatment, before this prednisolone regimen was repeated for another two cycles. Prednisolone treated men, who recovered from anti-sperm antibodies, underwent then sperm penetration assay (SPA) using zona-free hamster ova. Couples with male partners having negative SPA results (equal or less than five) were admitted to intracytoplasmic sperm injection (ICSI) cycles.
  Prednisolone treatment: Infertile men were treated with prednisolone tablet, which is an intermediate acting corticosteroid, po, for 21 days of their wife's menstrual cycles. Briefly, the prednisolone regimen was
Period: Overall Study
Arm/Group | Prednisolone Treated Men / Positive SPA / IVF | Prednisolone Treated Men / Negative SPA / ICSI | Control Men / Positive SPA / IVF | Control Men / Negative SPA / ICSI
Started | 67 | 74 | 47 | 53
Completed | 50 | 53 | 46 | 48
Not Completed | 17 | 21 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Clinical Data of Control Men Underwent IVF | The Clinical Data of Treated Men Underwent IVF | The Clinical Data of Control Men Underwent ICSI | The Clinical Data of Treated Men Underwent ICSI | Total
Number analyzed (Participants) | 46 | 50 | 48 | 53 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 50 | 48 | 53 | 197
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 36.2 (7.8) | 37.9 (5.8) | 34.5 (3.8) | 34.2 (2.9) | 35.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 46 | 50 | 48 | 53 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 46 | 50 | 48 | 53 | 197
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 46 | 50 | 48 | 53 | 197
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Iraq | 46 | 50 | 48 | 53 | 197

OUTCOME MEASURES:

1. Primary Outcome: Number of Control and Treated Participants With Successful Live Births Following Conventional IVF or ICSI Cycles
Description: Live birth rates in treated and control patients undergoing conventional IVF or ICSI cycles as determined by the sperm penetration assay (SPA) of hamster zone free ova
Time Frame: Nine months (pregnancy term) after the in vitro fertilization.
Measure: Number; unit: participants
Arm/Group | Prednisolone Treated Men / Positive SPA / IVF | Prednisolone Treated Men / Negative SPA / ICSI | Control Men / Positive SPA / IVF | Control Men / Negative SPA / ICSI
Number analyzed (Participants) | 50 | 53 | 46 | 48
participants | 18 | 13 | 8 | 9

ADVERSE EVENTS:
Time Frame: Infertile men with positive titer of ASA were treated with prednisolone tablet for 21 days of their wife's menstrual cycles and for three cycles. This made the total duration of treatment for each individual three months throughout an experiment duration window of 15 months, starting from October 2014 till March 2016.
Description: Adverse effects included infection, nausea, vomiting, diarrhea, headache, and hypertension.
Arm/Group | Prednisolone Treated Men / Positive SPA / IVF | Prednisolone Treated Men / Negative SPA / ICSI | Control Men / Positive SPA / IVF | Control Men / Negative SPA / ICSI
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/53 | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/53 | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 0/53 | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes